CLINICAL TRIAL: NCT01001234
Title: A Worldwide, Randomized, Double Blind, Placebo-Controlled, Parallel Group Clinical Trial to Evaluate the Safety and Efficacy of Rizatriptan for the Acute Treatment of Migraine in Children and Adolescents
Brief Title: A Study to Evaluate the Efficacy and Tolerability of Rizatriptan for Treatment of Acute Migraine in Children and Adolescents (MK-0462-082 AM7)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0462-082; 2009_679 (Other: Merck Registration Number); CTRI/2010/091/000407 (Other: CTRI)
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Results first posted 2012-05-08 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2022-02

CONDITIONS: Migraine, Acute
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Stage 1: rizatriptan (Experimental)
  Interventions: Drug: rizatriptan
- Stage 1: placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Stage 2: rizatriptan (Experimental)
  Interventions: Drug: rizatriptan
- Stage 2: placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rizatriptan — For participants randomized to rizatriptan in Stage 1: a single 5 or 10 mg rizatriptan orally disintegrating tablet (ODT) was to be taken within 30 minutes of onset of qualifying migraine (defined as a migraine of moderate or severe intensity).
  Rizatriptan dose administered was based on participant weight at Screening: those <40 kg received 5 mg tablet, those ≥40 kg received 10 mg tablet.
  Other Names: Maxalt; MK-0462
  Arms: Stage 1: rizatriptan
Drug: placebo — For participants randomized to placebo in Stage 1: a single placebo ODT was to be taken within 30 minutes of onset of qualifying migraine.
  Arms: Stage 1: placebo
Drug: rizatriptan — For participants randomized to rizatriptan in Stage 2 (must have taken placebo in Stage 1 and was Non-Responder [moderate or severe pain 15 minutes after dose] to be randomized at Stage 2): a single 5 or 10 mg rizatriptan ODT was to be taken approximately 15 minutes post Stage 1 dose, to treat same qualifying migraine treated in Stage 1.
  Rizatriptan dose administered was based on participant weight at Screening: those <40 kg received 5 mg tablet, those ≥40 kg received 10 mg tablet.
  Other Names: Maxalt; MK-0462
  Arms: Stage 2: rizatriptan
Drug: placebo — For participants randomized to placebo in Stage 2 (must have taken placebo in Stage 1 and was Non-Responder to be randomized at Stage 2) or allocated to placebo in Stage 2 (took rizatriptan in Stage 1 and was Non-Responder): a single placebo ODT was to be taken approximately 15 minutes post Stage 1 dose, to treat same qualifying migraine treated in Stage 1.
  Arms: Stage 2: placebo

SUMMARY:
This Clinical Trial evaluates the Safety and Efficacy of Rizatriptan for the Acute Treatment of Migraine in Children and Adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Patient weighs at least 20 kg (44 pounds)
* Patient has had a history of migraine with or without aura > 6 months with >= 1 to <= 8 moderate or severe migraine attacks per month in the 2 months prior to screening Visit 1
* Patient has a history of migraine defined by International Headache Society (IHS) migraine definitions
* Patient is willing to stay awake for at least 2 hours after administration of the first dose of study medication
* Patient has not experienced satisfactory relief from migraine pain with nonsteroidal anti-inflammatory drugs (NSAIDs) or N-acetyl-p-aminophenol (APAP) treatment
* The parent or guardian and patient agree to the patient's participation in the study as indicated by parental/guardian signature on the consent form and

patient assent

- For patients taking migraine prophylactic medication, treatment regimen is stable and has been taken for at least 3 months prior to Visit 1.

Exclusion Criteria:

* Patient is pregnant or breast-feeding, or is a female expecting to conceive within the projected duration of study participation
* Patient has a history of mild migraine attacks or migraines that resolve in less than 2 hours
* Patient has basilar or hemiplegic migraine headaches
* Patient has >15 headache-days per month OR has taken medication for acute

headache on more than 10 days per month in any of the 3 months prior to screening

* Patient has uncontrolled high blood pressure, uncontrolled diabetes, human immunodeficiency virus (HIV), any

cancer, or any other significant disease

* Patient has a history or clinical evidence of cardiovascular problems or stroke
* Patient has either demonstrated hypersensitivity to or experienced a serious

adverse event in response to rizatriptan

* Patient did not experience satisfactory relief from migraine pain to prior treatment with 2 or more adequate courses of 5-hydroxytryptamine 1 (5HT1) agonists
* Patient has a recent history (within the past year) or current evidence of drug or alcohol abuse or is a "recreational user" of illicit drugs
* Patient is currently taking monoamine oxidase inhibitors, methysergide, selective serotonin reuptake inhibitors (SSRIs) or serotonin norepinephrine reuptake inhibitors (SNRIs) or propranolol, and is unable to tolerate withdrawal of these medications for the intervals required
* Patient is currently participating or has participated in a study with an

investigational compound or device within 30 days of screening

- Patient is legally or mentally incapacitated.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1382 (Actual)
Dates: Start 2009-11-30 (Actual); Primary Completion 2011-04-21 (Actual); Study Completion 2011-04-21 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho TW, Pearlman E, Lewis D, Hamalainen M, Connor K, Michelson D, Zhang Y, Assaid C, Mozley LH, Strickler N, Bachman R, Mahoney E, Lines C, Hewitt DJ; Rizatriptan Protocol 082 Pediatric Migraine Study Group. Efficacy and tolerability of rizatriptan in pediatric migraineurs: results from a randomized, double-blind, placebo-controlled trial using a novel adaptive enrichment design. Cephalalgia. 2012 Jul;32(10):750-65. doi: 10.1177/0333102412451358. Epub 2012 Jun 18. PMID 22711898

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants randomized to double-blind study medication (Stage 1 - placebo or rizatriptan in a 20:1 ratio) at the Screening visit were given study drug and administration instructions. If a participant had not treated a qualifying migraine attack within up to 2-4 months, he/she may have been discontinued from the study
Groups:
- Placebo/NA: Stage 1 - Randomized to single placebo oral tablet to be taken within 30 minutes of onset of qualifying migraine / Stage 2 - If Stage 1 dose was taken and participant was Responder (mild or no pain 15 minutes after dose), no further study medication was to be administered.
- Rizatriptan/NA: Stage 1 - Randomized to single rizatriptan 5 or 10 mg oral tablet to be taken within 30 minutes of onset of qualifying migraine / Stage 2 - If Stage 1 dose was taken and participant was Responder (mild or no pain 15 minutes after dose), no further study medication was to be administered.
- Placebo/Rizatriptan: Stage 1 - Randomized to single placebo oral tablet to be taken within 30 minutes of onset of qualifying migraine / Stage 2 - If Stage 1 dose was taken and participant was Non-Responder (moderate or severe pain 15 minutes after dose), Stage 2 randomization was to occur and participants in this reporting group received single rizatriptan 5 or 10 mg oral tablet. Stage 2 dose was administered approximately 15 minutes post Stage 1 dose, to treat same qualifying migraine treated in Stage 1. Stage 2 randomization was in a ratio of 1:1 rizatriptan:placebo.
- Placebo/Placebo: Stage 1 - Randomized to single placebo oral tablet to be taken within 30 minutes of onset of qualifying migraine / Stage 2 - If Stage 1 dose was taken and participant was Non-Responder (moderate or severe pain 15 minutes after dose), Stage 2 randomization was to occur and participants in this reporting group received single placebo oral tablet. Stage 2 dose was administered approximately 15 minutes post Stage 1 dose, to treat same qualifying migraine treated in Stage 1. Stage 2 randomization was in a ratio of 1:1 rizatriptan:placebo.
- Rizatriptan/Placebo: Stage 1 - Randomized to single rizatriptan 5 or 10 mg oral tablet to be taken within 30 minutes of onset of qualifying migraine / Stage 2 - If Stage 1 dose was taken and participant was Non-Responder (moderate or severe pain 15 minutes after dose), allocated to receive single placebo oral tablet in Stage 2 to treat same qualifying migraine treated in Stage 1 (Stage 2 dose to be administered 15 minutes post Stage 1 dose).
Period: Overall Study
Arm/Group | Placebo/NA | Rizatriptan/NA | Placebo/Rizatriptan | Placebo/Placebo | Rizatriptan/Placebo
Started | 492 (Participants who were randomized to study drug) | 31 (Participants who were randomized to study drug) | 409 (Participants who were randomized to study drug) | 410 (Participants who were randomized to study drug) | 40 (Participants who were randomized to study drug)
Particpants Treated | 124 (Participants who took study drug in Stage 1 and/or Stage 2) | 8 (Participants who took study drug in Stage 1 and/or Stage 2) | 400 (Participants who took study drug in Stage 1 and/or Stage 2) | 405 (Participants who took study drug in Stage 1 and/or Stage 2) | 40 (Participants who took study drug in Stage 1 and/or Stage 2)
Participants Not Treated | 368 (Participants who did not take study drug) | 23 (Participants who did not take study drug) | 9 (Participants who did not take study drug) | 5 (Participants who did not take study drug) | 0 (Participants who did not take study drug)
Completed | 87 (Participants who took study drug in Stage 1 and/or Stage 2 and completed study) | 5 (Participants who took study drug in Stage 1 and/or Stage 2 and completed study) | 377 (Participants who took study drug in Stage 1 and/or Stage 2 and completed study) | 385 (Participants who took study drug in Stage 1 and/or Stage 2 and completed study) | 40 (Participants who took study drug in Stage 1 and/or Stage 2 and completed study)
Not Completed | 405 | 26 | 32 | 25 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 0 | 0
Not completed — Protocol Violation | 34 | 3 | 19 | 18 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Not Treated: Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Not Treated: Withdrawal by Subject | 23 | 2 | 2 | 0 | 0
Not completed — Not Treated: Protocol Violation | 3 | 0 | 0 | 0 | 0
Not completed — Not Treated: Lost to Follow-up | 53 | 4 | 7 | 5 | 0
Not completed — Not Treated: Pregnancy | 3 | 0 | 0 | 0 | 0
Not completed — Not Treated: Physician Decision | 37 | 4 | 0 | 0 | 0
Not completed — Not Treated: Lack of Qualifying Event | 248 | 13 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/NA | Rizatriptan/NA | Placebo/Rizatriptan | Placebo/Placebo | Rizatriptan/Placebo | Total
Number analyzed (Participants) | 124 | 8 | 400 | 405 | 40 | 977
Age, Continuous [Mean (Standard Deviation); unit: years] — Includes only participants who took study drug
  years | 12.7 (2.9) | 13.4 (2.1) | 13.0 (2.9) | 13.1 (2.9) | 13.1 (3.4) | 13.0 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Includes only participants who took study drug
  Participants
    Female | 61 | 4 | 227 | 238 | 20 | 550
    Male | 63 | 4 | 173 | 167 | 20 | 427

OUTCOME MEASURES:

1. Primary Outcome: Pain Freedom at 2 Hours Post Dose in Participants Between 12 and 17 Years of Age
Description: Pain intensity was assessed using a 5-Face Pain Scale ranging from 1=no pain to 5=very bad pain. Pain freedom was defined as a reduction in severity from a rating of 3, 4 or 5 (moderate or severe pain) at the Stage 2 baseline (15 minutes post Stage 1 dose) to a rating of 1 (no pain) at 2 hours post Stage 2 dose. Missing data were imputed by carrying forward the preceding Stage 2 pain intensity values. Missing Stage 2 baseline values were imputed by carrying forward the Stage 1 baseline value, if available.
Time Frame: 2 hours post Stage 2 dose
Population: Includes participants who did not respond to placebo in Stage 1, were randomized to and took Stage 2 study drug and had both Stage 2 baseline migraine severity (moderate or severe) and at least one post Stage 2 dose efficacy measurement prior to or including the 2 hour post dose time point. Those randomized to rizatriptan in Stage 1 were excluded.
Measure: Number; unit: participants
Groups:
- Rizatriptan: Participants randomized to rizatriptan in Stage 2
- Placebo: Participants randomized to placebo in Stage 2
Arm/Group | Rizatriptan | Placebo
Number analyzed (Participants) | 284 | 286
participants
  2-hour pain freedom | 87 [25.3 to 36.4] | 63 [17.4 to 27.3]
  No 2-hour pain freedom | 197 | 223
Statistical Analysis 1: Comparison: Rizatriptan vs Placebo; The comparison of rizatriptan versus placebo with respect to the primary outcome was conducted using a logistic regression model with factors for treatment, Stage 2 baseline pain severity (moderate or severe) and region (United States [US] or ex-US). Model-derived odds ratio and a two-sided p-value were provided. An odds ratio >1 is in favor of the rizatriptan group; Test type: Superiority or Other; p = 0.025, Regression, Logistic — The statistical significance level for the primary endpoint was α=0.0477, and had been adjusted to account for the interim sample size adjustment; Testing of primary endpoint and secondary endpoints was conducted sequentially in a pre-specified order, thus strongly controlling Type I error; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.06 to 2.26]

2. Secondary Outcome: Pain Relief at 2 Hours Post Dose in Participants Between 12 and 17 Years of Age
Description: Pain intensity was assessed using a 5-Face Pain Scale ranging from 1=no pain to 5=very bad pain. Pain relief was defined as a reduction in severity from a rating of 3, 4 or 5 (moderate or severe pain) at the Stage 2 baseline (15 minutes post Stage 1 dose) to a rating of 2 or 1 (mild or no pain) at 2 hours post Stage 2 dose. Missing data were imputed by carrying forward the preceding Stage 2 pain intensity values. Missing Stage 2 baseline values were imputed by carrying forward the Stage 1 baseline value, if available.
Time Frame: 2 hours post Stage 2 dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Rizatriptan | Placebo
Number analyzed (Participants) | 284 | 286
participants
  2-hour pain relief | 167 [52.8 to 64.6] | 147 [45.4 to 57.3]
  No 2-hour pain relief | 117 | 139
Statistical Analysis 1: Comparison: Rizatriptan vs Placebo; The comparison of rizatriptan versus placebo with respect to pain relief at 2 hours post Stage 2 dose for participants between 12 and 17 years of age was conducted using a logistic regression model with factors for treatment, Stage 2 baseline pain severity (moderate or severe) and region (US or ex-US). Model-derived odds ratio and a two-sided p-value were provided. An odds ratio >1 is in favor of the rizatriptan group; Test type: Superiority or Other; p = 0.080, Regression, Logistic — Secondary endpoints were to be formally tested only if the test of the primary endpoint was statistically significant at the α=0.0477 level. The secondary endpoints were then tested sequentially in a pre-specified order, each at the α=0.05 level; This first secondary hypothesis was not statistically significant, therefore the other two were not formally tested for statistical significance; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.96 to 1.90]

3. Secondary Outcome: Pain Freedom at 2 Hours Post Dose in Participants Between 6 and 17 Years of Age
Description: as for outcome 1
Time Frame: 2 hours post Stage 2 dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Rizatriptan | Placebo
Number analyzed (Participants) | 382 | 388
participants
  2-hour pain freedom | 126 [28.3 to 37.9] | 94 [20.0 to 28.8]
  No 2-hour pain freedom | 256 | 294
Statistical Analysis 1: Comparison: Rizatriptan vs Placebo; The comparison of rizatriptan versus placebo with respect to pain freedom at 2 hours post Stage 2 dose for participants between 6 and 17 years of age was conducted using a logistic regression model with factors for treatment, Stage 2 baseline pain severity (moderate or severe), age (6 to 11 years old or 12 to 17 years old), and region (US or ex-US). Model-derived odds ratio and a two-sided p-value were provided. An odds ratio >1 is in favor of the rizatriptan group; Test type: Superiority or Other; p = 0.010, Regression, Logistic — This second secondary hypothesis was not formally tested since the first secondary was not statistically significant; Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.10 to 2.10]

4. Secondary Outcome: Pain Relief at 2 Hours Post Dose in Participants Between 6 and 17 Years of Age
Description: as for outcome 2
Time Frame: 2 hours post Stage 2 dose
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Rizatriptan | Placebo
Number analyzed (Participants) | 382 | 388
participants
  2-hour pain relief | 220 [52.5 to 62.6] | 204 [47.5 to 57.6]
  No 2-hour pain relief | 162 | 184
Statistical Analysis 1: Comparison: Rizatriptan vs Placebo; The comparison of rizatriptan versus placebo with respect to pain relief at 2 hours post Stage 2 dose for participants between 6 and 17 years of age was conducted using a logistic regression model with factors for treatment, Stage 2 baseline pain severity (moderate or severe), age (6 to 11 years old or 12 to 17 years old), and region (US or ex-US). Model-derived odds ratio and a two-sided p-value were provided. An odds ratio >1 is in favor of the rizatriptan group; Test type: Superiority or Other; p = 0.178, Regression, Logistic — This third secondary hypothesis was not formally tested since the first secondary was not statistically significant; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.91 to 1.63]

ADVERSE EVENTS:
Time Frame: Up to 14 days post dose
Description: Includes all randomized participants who received at least one dose of study drug (i.e., participants who only took study drug in Stage 1 were also included). Participants were included in the treatment group corresponding to the study treatment they actually received, with active treatment taking precedence over placebo treatment.
Groups:
- Rizatriptan: Participants who took any rizatriptan during the study (Stage 1 or 2)
- Placebo: Participants who took only placebo during the study
Arm/Group | Rizatriptan | Placebo
Serious Adverse Events (participants affected / at risk) | 0/462 | 2/515
Other Adverse Events (participants affected / at risk) | 0/462 | 0/515
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rizatriptan (N=462) | Placebo (N=515)
Enterobacter bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator agrees to delay publication of study results until Food and Drug Administration (FDA) grants pediatric exclusivity on the study drug. Investigator may publish results for his/her study site after primary publication of results of entire multicenter trial. Sponsor must be able to review all proposed results communications regarding study 60 days prior to submission for publication/presentation. Information identified by the Sponsor as confidential must be deleted prior to submission.